CLINICAL TRIAL: NCT05534763
Title: Internet-delivered Emotion Regulation Treatment (I-ER GD) for Transgender Adults and Co-occurring Mental Health Problems
Brief Title: Internet-delivered Treatment for Transgender Individuals With Co-occurring Mental Health Problems
Acronym: IERGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Hanna Sahlin, Principal investigator, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-00577-01
Record Dates: First submitted 2022-08-30; First posted 2022-09-09 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Gender Dysphoria; Emotion Regulation; Internet Delivered Treatment
MeSH Terms: conditions — Gender Dysphoria; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Study 1 is a feasibility study with pre- and post-assessments evaluating feasibility, acceptability and satisfaction of the study protocol and the preliminary efficacy of I-ER. Study 1 consists of IERGD (a behavioral intervention for individuals with GD) and IER SUPPORT (a parallell behavioral course for a support person to the person with GD).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IERGD (Experimental): I-ER GD is a 10-week intervention directed to the person with GD, provided via the internet with therapist-support. During treatment, participants have an assigned psychologist to interact with and be offered support by, either through feedback on assignments, asynchronous chats or, if needed, by telephone. I-ER GD will focus on increasing adaptive emotion regulation skills, healthy identity development, interpersonal effectiveness skills, coping and building a resilient lifestyle through psychoeducation on gender minority stress, practicing adaptive emotion regulation skills, and reducing emotional and behavioral avoidance.
  Interventions: Behavioral: IERGD
- IER SUPPORT (Other): I-ER Support is a 5-week intervention directed to a support person, provided as an optional addition to I-ER GD. I-ER Support is administered in the same manner and in parallel to the I-ER GD intervention. Treatment content is based on the same principles as I-ER GD, but from the perspective of increasing emotional support and understanding of GD. The support person could benefit from increased coping and emotion regulation skills, as they may also be exposed to discrimination or stigma due to having a transgender child, sibling or loved one. In better understanding the processes of being stigmatized and with improved emotion regulation skills, the support person may offer better support and help alleviate burdening effects for the individual with GD. For this reason, I-ER support is primarily aimed at people without trans-experience.
  Interventions: Other: IER SUPPORT

INTERVENTIONS:
Behavioral: IERGD — A 10 week behavioral treatment focusing on gender minority stress, maladaptive and adaptive emotion regulation, emotional awareness, the functionality of emotions, interpersonal skills and values and valued actions.
  Arms: IERGD
Other: IER SUPPORT — A 5-week behavioral course for a designated support person (family, friend, other) to the person with GD. The course focuses on teachings on living with minority stress, maladaptive and adaptive emotion regulation, emotional awareness, validation, interpersonal skills and values.
  Arms: IER SUPPORT

SUMMARY:
This project aims to develop and evaluate if an internet delivered psychological intervention for transgender individuals undergoing assessment for gender dysphoria and a support person, is feasible, acceptable and effective in increasing emotional skills, strengthening a healthy identity development, social support and resilience to current and future mental illness.

In two studies, a psychological treatment for transgender adults (18+) seeking health care for gender dysphoria and a support person (i.e., relative, friend) will be evaluated.

The project will be carried out at a specialized unit for transgender health care (ANOVA) at Karolinska University Hospital

DETAILED DESCRIPTION:
There are no psychosocial treatments for young transgender adults seeking treatment for gender dysphoria - psychological distress due to the incongruence between one's assigned sex and one's gender identity. This project aims to develop and evaluate if an internet delivered psychological intervention for individuals undergoing assessment for gender dysphoria and a support person, is feasible, acceptable and effective in increasing emotional skills, strengthening a healthy identity development, social support and resilience to current and future mental illness.

Data and Method: In three studies, a psychological treatment for transgender adults (18+) seeking care for gender dysphoria and a support person (i.e., relative, friend) will be evaluated. Study 1 is a feasibility study (N=40) with pre-, post- and weekly assessments evaluating the intervention's feasibility, credibility, acceptability and preliminary efficacy. Study 2 is a qualitative interview study exploring participants' experience of the intervention.

Plan for project realization: The project will be carried out at a specialized unit for transgender health care (ANOVA) at Karolinska University Hospital, with a large patient recruitment base and extensive experience of clinical studies providing good opportunities for later implementation in regular care.

Relevance: Studies show elevated rates of psychopathology in transgender adults. It has been suggested that experiences of minority stress, e.g., discrimination, internalized transphobia and gender identity concealment exhausts the ability to regulate negative emotions in an adaptive way. There is a need for treatment and preventive psychological interventions, particularly as the number of young transgender adults seeking gender affirming treatment has increased markedly during the 2000s. This project will lead to increased knowledge about the specific needs of this growing patient group and develop health care in accordance with national guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having had an initial assessment at ANOVA for GD between March 2022 and November 2022 and found eligible for a diagnostic assessment period and having been put on a waitlist for continued evaluation.
2. Being at least 18 years of age;
3. Reporting elevated self-perceived psychiatric symptoms (e.g., depression, anxiety, suicidality) or functional impairment (difficulties maintaining school, work or daily routines);
4. Be able to write and read in Swedish; and
5. Have daily access to a computer with internet connection.

Exclusion Criteria:

1. Evidence of active untreated mania, psychosis or other severe psychiatric symptoms that are deemed primary and need treatment;
2. Current and increased suicide risk, such as intrusive suicide thoughts, or current suicide plans, or recent suicide attempt;
3. Current enrollment in another psychological intervention study or currently receiving regular psychological treatment or
4. Less than 6 weeks of stable psychopharmacotherapy if such treatment is ongoing.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited to I-ER GD. | At pretreatment.
  Measures will include recruitment rate during study inclusion period (0-30 participants).
Client Satisfaction Questionnaire (CSQ-8; Attkisson & Zwick, 1982) in I-ER GD | At post-treatment (week 12).
  Measures treatment satisfaction after treatment. Range 8-32, higher values equals higher satisfaction with treatment.
The Credibility and Expectancy Questionnaire (Devilly & Borkovec, 2000) in I-ER GD. | At treatment week 2.
  Measures treatment credibility and expectancy for positive change. Range 0-5, higher values equals higher treatment credibility and expectancy.
The Negative effects Questionnaire (NEQ; Rozental et al. 2016) in I-ER GD. | At post-treatment (week 12).
  Measures negative effects of psychological treatment after an intervention. Range 0-20, higher values equals worse outcomes, and more negative effects of treatment.
The internet intervention Patient Adherence Scale (iiPAS; Lenhard et al. 2019) in I-ER GD | At mid-treatment (week 5).
  Measures adherence to treatment at two timepoints of the treatment. Range 0-20. Higher scores indicate better adherence.
The internet intervention Patient Adherence Scale (iiPAS; Lenhard et al. 2019) in I-ER GD | At post-treatment (week 12).
  Measures adherence to treatment at two timepoints of the treatment. Range 0-20. Higher scores indicate better adherence.
Number of participants recruited to I-ER SUPPORT. | At pretreatment.
  Measures will include recruitment rate during study inclusion period (0-15 participants).
The Client Satisfaction Questionnaire (CSQ-8; Attkisson & Zwick, 1982) in I-ER SUPPORT | At post-treatment (week 10).
  Measures treatment satisfaction. Range 8-32, higher values equals higher satisfaction with treatment.
The Credibility and Expectancy Questionnaire (Devilly & Borkovec, 2000) in I-ER SUPPORT | At treatment week 2.
  Measures treatment credibility and expectancy for positive change. Range 0-5, higher values equals higher treatment credibility and expectancy.
The Negative effects Questionnaire (NEQ; Rozental et al. 2016) in I-ER SUPPORT. | At post-treatment (week 10).
  Measures negative effects of psychological treatment. Range 0-20, higher values equals worse outcomes, and more negative effects of treatment.

SECONDARY OUTCOMES:
Changes in Gender minority stress and resilience (GMSR, Testa et al 2014) for I-ER GD. | At pre-treatment and at post treatment (week 12)
  Changes in the Gender minority stress and resilience scale. Range 0-17 for sub scales Gender related discrimination, rejection, victimization. Higher values represents higher levels of discrimination, rejection, victimization etc. Range 0-164 for sub scales Non-affirmation of gender identity, Internalized transphobia, Pride, Negative expectations for the future, Nondisclosure and Community connectedness. Higher values represents higher levels of whatever the sub scale covers (e.g. pride, internalized transphobia, community connectedness etc).
Changes in The Difficulties in emotion regulation scale, (DERS-16; Gratz & Roemer, 2004) for I-ER GD. | At pre-treatment and at post treatment (week 12)
  Changes in the Difficulties in emotion regulation scale, DERS-16. Range 16-80. Lower values equals better outcomes.
Changes in The Difficulties in emotion regulation scale, (DERS-16; Gratz & Roemer, 2004) for I-ER GD. | Weekly during the treatment (weeks 1-11)
  Changes in the Difficulties in emotion regulation scale, DERS-16. Range 16-80. Lower values equals better outcomes.
Changes in The Emotion Regulation Questionnaire, (ERQ; Gross & John, 2003) for I-ER GD. | At pre-treatment and at post treatment (week 12)
  Changes in the Emotion Regulation Questionnaire, ERQ. Subscales Cognitive reappraisal (Range 6-42). and Suppression (Range 4-28). Higher values equals better outcomes in reappraisal, and worse outcomes in Suppression.
Changes inThe Alcohol Use Disorders Identification Test (AUDIT; Berman, Wennberg & Källmén, 2012) for I-ER GD. | At baseline and at post treatment (week 12)
  Changes in alcohol consumption. Range 0-40 where higher values equal higher substance use, worse outcomes.
Changes inThe Drug Use Disorders Identification Test (DUDIT; Berman, Wennberg & Källmén, 2012) for I-ER GD. | At baseline and at post treatment (week 12)
  Changes in drug consumption. Range 0-44 where higher values equal higher substance use, worse outcomes.
Changes in Gender Congruence and Life Satisfaction Scale (GCLS; Dhejne et al. 2019) for I-ER GD | At baseline and at post treatment (week 12)
  Change and measure improvements in gender (in)congruence, related mental well-being, and life satisfaction throughout the process of undergoing gender affirming medical interventions. Range: 38-190 where higher values indicate greater gender congruence, greater gender-related well-being, and greater life satisfaction.
Changes in Work and social adjustment scale (WSAS; Marks 1986) for I-ER GD | At baseline and at post treatment (week 12)
  Changes in functioning. Ranges from 0-40 where higher scores indicate a more impaired functioning.
Changes in Social Interaction Anxiety Scale (SIAS; Mattick & Clarke 1998) for I-ER GD | At pre-treatment and at post treatment (week 12)
  Changes in anxiety over 20 different situations. Ranges from 0-80 where higher scores indicate a higher social anxiety.
Changes in Social Interaction Anxiety Scale (SIAS; Mattick & Clarke 1998) for I-ER GD | Weekly during the treatment (weeks 1-11)
  Changes in anxiety over 20 different situations. Ranges from 0-80 where higher scores indicate a higher social anxiety.
Changes in Montgomery Åsberg Depression Rating Scale (MADRS-S; Montgomery & Åsberg 1979) for I-ER GD | At pre-treatment and post treatment (week 12)
  Changes in depressive symptoms. Ranges from 0-54 where higher scores indicate higher depressive severity.
Changes in Deliberate Self-Harm Inventory (DSHI-9; Lundh, Karim & Quillisch 2007) for I-ER GD | At pre-treatment and at post treatment (week 12)
  Changes in instances and forms of self-harming behavior. Higher number of instances indicates worse outcomes.
Changes in Deliberate Self-Harm Inventory (DSHI-9; Lundh, Karim & Quillisch 2007) for I-ER GD | Weekly during the treatment (weeks 1-11)
  Changes in instances and forms of self-harming behavior. Higher number of instances indicates worse outcomes.
Changes in Brunnsviken Brief Quality of Life Inventory (BBQ; Lindner et al, 2016) for I-ER GD | At pre-treatment and at post treatment (week 12)
  Changes in perceived quality of life. Range: 0-96. Higher scores indicate a higher perceived quality of life.
Changes in Satisfaction With Life, Swedish (SWLS; Diener 1985) for I-ER GD | At pre-treatment and at post treatment (week 12)
  Changes in global cognitive judgements of one's life. Range: 0-35. Higher score indicates higher satisfaction with one's life.
Changes in Perceived Stress Scale (PSS-14; Cohen, Kamarck & Mermelstein 1983) for I-ER GD | At pre-treatment and at post treatment (week 12)
  Changes in perceived stress. Range: 0-56. Higher scores indicate greater perceived stress.
Changes in Multidimensional Scale of Perceived Social Support (MSPSS; Zimet et al, 1988) for I-ER GD | At pre-treatment and at post treatment (week 12)
  Changes in perceived support from family, friends and significant other(s). Range: 12-84. Higher scores indicate greater perceived stress.
Changes in Rosenberg's scale of self-esteem (Rosenberg; Schmitt & Allik 2005) for I-ER GD | At pre-treatment and at post treatment (week 12)
  Changes in self-esteem. Range: 0-40. Higher scores indicate higher self-esteem.
Changes in Rumination Response Scale (RRS-10; Nolen-Hoeksema, Morrow 1991) for I-ER GD | At pre-treatment and at post treatment (week 12)
  Changes in ruminative tendencies. Range: 10-40. Higher scores indicate higher levels of ruminative response styles.
Changes in Affect Labeling Questionnaire (ALQ; Sahi et al, in prep.) for I-ER GD | At pre-treatment and at post treatment (week 12)
  Changes in one's ability to recognize emotions. Range 12-60. Higher scores indicates higher ability to recognize and label emotions.
Changes in The Gender/Sex diversity belief scale (GSDB; Schudson & van Anders, 2022) for I-ER SUPPORT | At pre-treatment and at post treatment (week 10)
  Changes in the Gender/Sex diversity belief scale. Range 23-161. Higher values equals more positive attitudes toward transgender individuals.
Changes in Affect Labeling Questionnaire (ALQ; Sahi et al, in prep.) for I-ER SUPPORT | At pre-treatment and at post treatment (week 10)
  Changes in one's ability to recognize emotions. Range 12-60. Higher scores indicates higher ability to recognize and label emotions.
Changes in The Emotion Regulation Questionnaire, (ERQ; Gross & John, 2003) for I-ER SUPPORT. | At pre-treatment and at post treatment (week 10)
  Changes in the Emotion Regulation Questionnaire, ERQ. Subscales Cognitive reappraisal (Range 6-42). and Suppression (Range 4-28). Higher values equals better outcomes in reappraisal, and worse outcomes in Suppression.
Changes in The Difficulties in emotion regulation scale, (DERS-16; Gratz & Roemer, 2004) for I-ER SUPPORT | At pre-treatment and at post treatment (week 10)
  Changes in the Difficulties in emotion regulation scale, DERS-16. Range 16-80. Lower values equals better outcomes.
Changes in The Difficulties in emotion regulation scale, (DERS-16; Gratz & Roemer, 2004) for I-ER SUPPORT | Weekly during the treatment (weeks 1-10)
  Changes in the Difficulties in emotion regulation scale, DERS-16. Range 16-80. Lower values equals better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Sahlin, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- ANOVA, Karolinska University Hospital, Norra Stationsgatan 69, Plan 4, Stockholm, Sweden